CLINICAL TRIAL: NCT00014989
Title: Randomized Clinical Trial of the Beneficial Effects of Antenatal Magnesium Sulfate (BEAM)
Brief Title: Beneficial Effects of Antenatal Magnesium Sulfate (BEAM Trial)
Acronym: BEAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: NICHD-0800; U10HD021414 (NIH); U10HD021410 (NIH); U10HD027905 (NIH); U10HD027917 (NIH); U10HD027860 (NIH); U10HD027915 (NIH); U10HD034116 (NIH); U10HD034208 (NIH); U10HD034136 (NIH); U10HD027869 (NIH); U10HD036801 (NIH); U10HD027861 (NIH); U10HD034122 (NIH); U10HD034210 (NIH); U10HD040500 (NIH); U10HD040485 (NIH); U10HD053097 (NIH); U10HD040544 (NIH); U10HD040545 (NIH); U10HD040560 (NIH); U10HD040512 (NIH)
Record Dates: First submitted 2001-04-17; First posted 2001-04-18 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Cerebral Palsy; Intraventricular Hemorrhage; Periventricular Leukomalacia; Pulmonary Edema; Abruptio Placentae
Keywords: Preterm delivery; Cerebral palsy; Magnesium sulfate
MeSH Terms: conditions — Cerebral Palsy; Leukomalacia, Periventricular; Pulmonary Edema; Abruptio Placentae; Premature Birth | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: magnesium sulfate

SUMMARY:
As many more premature infants survive, the numbers of these infants with health problems increases. The rate of cerebral palsy (CP) in extremely premature infants is approximately 20%. Magnesium sulfate, the most commonly used drug in the US to stop premature labor, may prevent CP. This trial tests whether magnesium sulfate given to a woman in labor with a premature fetus (24 to 31 weeks out of 40) will reduce the rate of death or moderate to severe CP in the children at 2 years. The children receive ultrasounds of their brains as infants and attend three follow-up visits over two years to assess their health and development.

DETAILED DESCRIPTION:
The prevalence of cerebral palsy is increasing as the survival rate of extremely premature infants is improving. Studies have suggested an apparent association between maternal magnesium sulfate administration and a reduced risk of cerebral palsy. Other studies have suggested a possible association between magnesium sulfate and a reduction in neonatal cranial ultrasound abnormalities which may be markers for subsequent development of cerebral palsy.

This multicenter trial tests whether prophylactic magnesium sulfate given to women, for whom preterm delivery is imminent, reduces the risk of death or moderate to severe cerebral palsy in their children. Women presenting from 24.0 to 31.6 weeks gestation with advanced preterm labor or premature rupture of the membranes (pPROM) and no recent exposure to magnesium sulfate are randomized to receive either intravenous magnesium sulfate or masked study drug placebo. The study drug is administered as a 6 gram loading dose followed by a 2 gram/hour infusion (or equivalent rate for placebo). If after 12 hours, delivery has not occurred and is not anticipated, the infusion is stopped. No other parenteral tocolytics other than the IV medication may be used. Retreatment with study medication is given any time labor recurs or delivery is anticipated until gestational age is > 34.0 wks. Standard clinical management and therapy is to be maintained for all study patients. Patients are assessed for signs of intolerance to the study medications and maternal data are collected up to hospital discharge. A sample of venous blood is collected and neonatal cranial ultrasounds are performed. Up to three follow-up visits are scheduled over two years where certified examiners, masked to study group assignment, collect physical and neurological data, including a modified Gross Motor Function Classification Scale. The Bayley Scales of Infant Development is also administered. Cranial ultrasounds are reviewed centrally.

The primary outcome is a composite outcome of death or moderate to severe cerebral palsy. Secondary outcomes include maternal infectious morbidity, pulmonary edema and placental abruption, neonatal stillbirth and death, intraventricular hemorrhage, periventricular leukomalacia, neonatal infectious and noninfectious morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant with diagnosis of preterm labor
* Membrane rupture or delivery definitely planned within 24 hours
* Gestational age > 24.0 and < 31.6 wks, viable fetus

Exclusion Criteria:

* Prior IV magnesium sulfate therapy within 12 hours of screening
* Delivery expected <2 hrs
* Cervical dilation > 8 cm
* More than 2 fetuses
* Known major fetal anomalies
* Hypertension or preeclampsia
* Maternal medical complications contraindicating magnesium sulfate treatment
* Participation in any intervention study which influences infant neurological outcome
* Previous participation in this trial

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2136 (Actual)
Dates: Start 1997-12; Primary Completion 2007-02 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Composite outcome of death or moderate to severe cerebral palsy

SECONDARY OUTCOMES:
Maternal
Chorioamnionitis
Endometritis
Other infectious morbidity
Pulmonary edema
Placental abruption
Neonatal
Stillbirth and neonatal death
Intraventricular hemorrhage
Neonatal infectious morbidity
Neonatal noninfectious morbidity
Birth weight
Days in NICU

CONTACTS AND LOCATIONS:
Overall Officials: Dwight Rouse, MD, Principal Investigator — University of Alabama at Birmingham; Menachem Miodovnik, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (17):
- United States (17):
  - University of Alabama, Birmingham, Alabama
  - Dept of OB/GYN, University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Dept of OB/GYN, Hutzel Hospital, Detroit, Michigan
  - St. Luke's - Roosevelt Hospital, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Forsyth Memorial Hospital, Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - The University Hospital, University of Cincinnati, Cincinnati, Ohio
  - Case Western University, Cleveland, Ohio
  - Dept of OB/GYN, Ohio State University, Columbus, Ohio
  - MCP Hahnemann University, Philadelphia, Pennsylvania
  - Dept of OB/GYN Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Dept of OB/GYN, Southwestern Medical Center, University of Texas, Dallas, Texas
  - University of Texas Medical Branch - Galveston, Galveston, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared after completion and publication of the main analyses in accordance with NIH policy. The dataset can be obtained by email at mfmudatasets@bsc.gwu.edu.

REFERENCES:
- [Background] Nelson KB, Grether JK. Can magnesium sulfate reduce the risk of cerebral palsy in very low birthweight infants? Pediatrics. 1995 Feb;95(2):263-9. PMID 7838646
- [Background] Schendel DE, Berg CJ, Yeargin-Allsopp M, Boyle CA, Decoufle P. Prenatal magnesium sulfate exposure and the risk for cerebral palsy or mental retardation among very low-birth-weight children aged 3 to 5 years. JAMA. 1996 Dec 11;276(22):1805-10. PMID 8946900
- [Background] Hallak M, Berry SM, Madincea F, Romero R, Evans MI, Cotton DB. Fetal serum and amniotic fluid magnesium concentrations with maternal treatment. Obstet Gynecol. 1993 Feb;81(2):185-8. PMID 8423946
- [Background] Aziz K, Vickar DB, Sauve RS, Etches PC, Pain KS, Robertson CM. Province-based study of neurologic disability of children weighing 500 through 1249 grams at birth in relation to neonatal cerebral ultrasound findings. Pediatrics. 1995 Jun;95(6):837-44. PMID 7761206
- [Background] Pinto-Martin JA, Riolo S, Cnaan A, Holzman C, Susser MW, Paneth N. Cranial ultrasound prediction of disabling and nondisabling cerebral palsy at age two in a low birth weight population. Pediatrics. 1995 Feb;95(2):249-54. PMID 7838643
- [Result] Rouse DJ, Hirtz DG, Thom E, Varner MW, Spong CY, Mercer BM, Iams JD, Wapner RJ, Sorokin Y, Alexander JM, Harper M, Thorp JM Jr, Ramin SM, Malone FD, Carpenter M, Miodovnik M, Moawad A, O'Sullivan MJ, Peaceman AM, Hankins GD, Langer O, Caritis SN, Roberts JM, for the Eunice Kennedy Shriver NICHD Maternal-Fetal Medicine Units Network. A randomized, controlled trial of magnesium sulfate for the prevention of cerebral palsy. New England Journal of Medicine, 359:895-905, 2008.
- [Result] Costantine MM, Weiner SJ; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units Network (MFMU). Effects of antenatal exposure to magnesium sulfate on neuroprotection and mortality in preterm infants: a meta-analysis. Obstet Gynecol. 2009 Aug;114(2 Pt 1):354-364. doi: 10.1097/AOG.0b013e3181ae98c2. PMID 19622997
- [Derived] Buhimschi CS, Jablonski KA, Rouse DJ, Varner MW, Reddy UM, Mercer BM, Leveno KJ, Wapner RJ, Sorokin Y, Thorp JM Jr, Ramin SM, Malone FD, Carpenter MW, O'Sullivan MJ, Peaceman AM, Saade GR, Dudley D, Caritis SN, Buhimschi IA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Cord Blood Haptoglobin, Cerebral Palsy and Death in Infants of Women at Risk for Preterm Birth: A Secondary Analysis of a Randomised Controlled Trial. EClinicalMedicine. 2019 Mar 22;9:11-18. doi: 10.1016/j.eclinm.2019.03.009. eCollection 2019 Mar. PMID 31143877
- [Derived] Hirtz DG, Weiner SJ, Bulas D, DiPietro M, Seibert J, Rouse DJ, Mercer BM, Varner MW, Reddy UM, Iams JD, Wapner RJ, Sorokin Y, Thorp JM Jr, Ramin SM, Malone FD, Carpenter MW, O'Sullivan MJ, Peaceman AM, Hankins GD, Dudley D, Caritis SN; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Antenatal Magnesium and Cerebral Palsy in Preterm Infants. J Pediatr. 2015 Oct;167(4):834-839.e3. doi: 10.1016/j.jpeds.2015.06.067. Epub 2015 Aug 5. PMID 26254839
- [Derived] Twickler DM, McIntire DD, Alexander JM, Leveno KJ. Effects of magnesium sulfate on preterm fetal cerebral blood flow using Doppler analysis: a randomized controlled trial. Obstet Gynecol. 2010 Jan;115(1):21-25. doi: 10.1097/AOG.0b013e3181c4f7c1. PMID 20027029
- [Derived] Rouse DJ, Hirtz DG, Thom E, Varner MW, Spong CY, Mercer BM, Iams JD, Wapner RJ, Sorokin Y, Alexander JM, Harper M, Thorp JM Jr, Ramin SM, Malone FD, Carpenter M, Miodovnik M, Moawad A, O'Sullivan MJ, Peaceman AM, Hankins GD, Langer O, Caritis SN, Roberts JM; Eunice Kennedy Shriver NICHD Maternal-Fetal Medicine Units Network. A randomized, controlled trial of magnesium sulfate for the prevention of cerebral palsy. N Engl J Med. 2008 Aug 28;359(9):895-905. doi: 10.1056/NEJMoa0801187. PMID 18753646
- See also: Click here for more information on the NICHD MFMU Research Network. — http://www.bsc.gwu.edu/mfmu/